CLINICAL TRIAL: NCT06004531
Title: Planetary Health and Loneliness: Survey and Mini-intervention to Study the Interrelations of Multiple Behavior Change and Perception of Social Isolation
Brief Title: Planetary Health and Loneliness
Acronym: PAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs University Bremen gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CUB_PHAL2023; Lippke202308 (Other: Constructor University (formerly Jacobs University))
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Loneliness; Anxiety; Health-Related Behavior; Healthy Lifestyle; Healthy Nutrition; Healthy Diet; Health Behavior
Keywords: Planetary Health; Eco-Friendly Behavior; Eco-Anxiety; Covid-19
MeSH Terms: conditions — Anxiety Disorders; Health Behavior; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Promoting (Experimental): The survey will be organized so health promoting behavioral scale questions will be asked first concerning personal wellbeing. This will be followed by eco-friendly behavior scale questions involving one's concern for the wellbeing of the planet. After this, there will be two surveys concerning loneliness and eco-anxiety before the intervention.
  Interventions: Behavioral: Prompting open-ended question promoting sustainability; Behavioral: Sustainability Passage
- Eco-friendly behavior (Experimental): The survey will be organized so eco-friendly behavior scale questions involving one's concern for the wellbeing of the planet will be asked first. This will be followed by health promoting behavioral scale questions concerning personal wellbeing. After this, there will be two surveys concerning loneliness and eco-anxiety before the intervention.
  Interventions: Behavioral: Prompting open-ended question promoting sustainability; Behavioral: Sustainability Passage

INTERVENTIONS:
Behavioral: Prompting open-ended question promoting sustainability — This intervention will include active persuasion through prompting participants to answer an open-ended question regarding how they will alter their behavior to become more sustainable and eco-friendly.
Behavioral: Sustainability Passage — This intervention will include passive persuasion through presenting participants with a passage discussing the serious issue of climate change and the pressing need for systemic and individual change to adopt sustainable practices and lifestyles.

SUMMARY:
The aim of this online study is the evaluation of planetary health behaviors in relation to levels of eco-anxiety, general well-being, and levels of loneliness. As climate change progresses at a dangerous rate, it is important to establish and maintain lifestyles that are productive, fulfilling, environmentally conscious, and low in anxiety. Through a better understanding of the interconnected nature of planetary health behaviors with other aspects of healthy living and perception of social isolation, this study will add to current state of science to help inform the creation of interventions promoting sustainable, healthy, happy living among the general public and specific subgroups.

DETAILED DESCRIPTION:
The aim of this online study is the evaluation of healthy behaviors and anxiety levels in relation to selected physical, mental, and environmental health aspects. The umbrella terminology of "planetary health" is used in the context of this study. As climate change progresses at a dangerous rate, it is important to establish and maintain lifestyles that are productive, fulfilling, environmentally conscious, and low in anxiety. By evaluating prevalence of healthy behaviors and levels of eco-anxiety as well as loneliness as one early indicator of health risk, this study hopes to build on existing public health knowledge to develop interventions targeting and encouraging multiple aspects of healthy, eco-friendly lifestyles. This study will also help later intervention design by determining effective methods of persuasion and promotion of sustainable planetary health behaviors. Main research questions are

I. Are climate-sensitive people and rehabilitation patients (in terms of EMCB, YCSCB and Mindful Health) more likely to also promote their own health (in terms of physical activity and healthy nutrition)? II. What is the (non-)linear relationship between eco-anxiety and climate-sensitiveness/health behavior? III. Is climate-sensitiveness and eco-anxiety invariant to partner status, number of people in the household, gender, occupation, and age? (No differences) IV. Is loneliness linked to partner status, number of people in the household and younger age but uncorrelated to eco-anxiety, climate-sensitiveness/health behavior? V. What is the prevalence of loneliness in 2023 in comparison to 2022, 2021, 2020, and 2019? Do people and rehabilitation patients who feel more lonely after the corona pandemic than before show more eco-anxiety and climate-sensitiveness but less healthy behavior than people who feel as/less lonely than prior to the corona pandemic? VI. Is active persuasion involving mental simulation more effective in promoting eco-friendly behaviours than passive persuasion involving information dissemination as measured by the YCSCB and EMCB? (testing two mini interventions) VII. To what extent are medical rehabilitation patients different from the general population?

ELIGIBILITY:
Inclusion Criteria:

* Ability to participate in surveys (e.g., sufficient German or English language skills)

Exclusion Criteria:

* Not being of age
* Illiteracy
* Massively limited cognitive abilities (linguistic components of the digital offerings must be able to be used and questionnaires completed or interviews participated in)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1684 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Young Consumers' Sustainable Consumption Behaviors (YCSCB) validated scale | This scale will take approximately 2 minutes to fill out completely.
  The primary outcome measure will be the YCSCB validated scale questionnaire. This will be given to participants right after they have completed the intervention section of the survey.
  The answering options range from "Never" (0, minimum score) to "Sometimes" (1) and "Often" (2) up to "Always" (3, maximum score). The items are worded
  1. I eat meat (steak, ham, etc.).
  2. I eat dairy products (butter, cheese, yoghurt, etc.).
  3. I keep a healthy diet.
  4. There are times when I discard food products.
  5. I buy locally grown food products.
  6. I reuse my leftovers for the next meal. and items # 1, 2 and 4 need to be reversed, then all items can be used as single items or as aggregated scales, with higher scores indicating a better outcome in terms of planetary health.
Ethically Minded Consumer Behavior (EMCB) validated scale | This scale will take approximately 2 minutes to fill out completely.
  The second primary outcome measure will be the EMCB validated scale questionnaire. This will be given to participants right after they have completed the intervention section of the survey.
  The answering options range from "Never true" (0, minimum score) to "Rarely true" (1), "Sometimes true" (2), "Mostly true" (3) and "Always true" (4, maximum score). The items are worded (for instance) 1. When there is a choice, I always choose the product that contributes to the least amount of environmental damage.
  2. I have switched products for environmental reasons. 3. If I understand the potential damage to the environment that some products can cause, I do not purchase those products.
  ... 10. I have paid more for socially responsible products when there is a cheaper alternative.
  All items can be used as single items or as aggregated scales, with higher scores indicating a better outcome in terms of planetary health.
Loneliness item from the Center for Epidemiological Studies-Depression-(CES D)-Scale | This item will take less than 1 minute to complete.
  To study some of the research questions unrelated to the intervention, the perceived social isolation is measured with a standardized scale building on the item in the Center for Epidemiological Studies-Depression-(CES-D)-Scale. The item is worded "How often did you feel lonely?" with the answering options "Daily" (3), "Several times a week" (2), "Once a week" (1) and "Rarely/never" (0).
  The item can be used as single items, with higher scores indicating a worse outcome in terms of more loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Dr., Principal Investigator — Constructor University
Locations (1):
- Germany, Bremen, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be published. Other researchers are welcome to get in contact with the PI to get access to anonymous data.

REFERENCES:
- [Background] Arias, P., Bellouin, N., Coppola, E., Jones, C., Krinner, G., Marotzke, J., Naik, V., Plattner, G.-K., Rojas, M., Sillmann, J., Storelvmo, T., Thorne, P., Trewin, B., Achutarao, K., Adhikary, B., Armour, K., Bala, G., Barimalala, R., Berger, S., & Zickfeld, K. (2021, January). Climate Change 2021: The Physical Science Basis. Contribution of Working Group I to the Sixth Assessment Report of the Intergovernmental Panel on Climate Change; Technical Summary.
- [Background] Bull ER, McCleary N, Li X, Dombrowski SU, Dusseldorp E, Johnston M. Interventions to Promote Healthy Eating, Physical Activity and Smoking in Low-Income Groups: a Systematic Review with Meta-Analysis of Behavior Change Techniques and Delivery/Context. Int J Behav Med. 2018 Dec;25(6):605-616. doi: 10.1007/s12529-018-9734-z. PMID 30003476
- [Background] Cheng J, Xu Z, Bambrick H, Prescott V, Wang N, Zhang Y, Su H, Tong S, Hu W. Cardiorespiratory effects of heatwaves: A systematic review and meta-analysis of global epidemiological evidence. Environ Res. 2019 Oct;177:108610. doi: 10.1016/j.envres.2019.108610. Epub 2019 Jul 26. PMID 31376629
- [Background] Dohle S, Hofmann W. Consistency and Balancing in Everyday Health Behaviour: An Ecological Momentary Assessment Approach. Appl Psychol Health Well Being. 2019 Mar;11(1):148-169. doi: 10.1111/aphw.12148. Epub 2018 Nov 13. PMID 30426704
- [Background] Druckman, A., & Jackson, T. (2016). Understanding Households as Drivers of Carbon Emissions. In R. Clift & A. Druckman (Eds.), Taking Stock of Industrial Ecology (pp. 181-203). Springer International Publishing. https://doi.org/10.1007/978-3-319-20571-7_9
- [Background] Ford ES, Bergmann MM, Boeing H, Li C, Capewell S. Healthy lifestyle behaviors and all-cause mortality among adults in the United States. Prev Med. 2012 Jul;55(1):23-7. doi: 10.1016/j.ypmed.2012.04.016. Epub 2012 Apr 29. PMID 22564893
- [Background] Geller K, Lippke S, Nigg CR. Future directions of multiple behavior change research. J Behav Med. 2017 Feb;40(1):194-202. doi: 10.1007/s10865-016-9809-8. Epub 2016 Oct 26. PMID 27785652
- [Background] Lacroix, K. (2018). Comparing the relative mitigation potential of individual pro-environmental behaviors. Journal of Cleaner Production, 195, 1398-1407. https://doi.org/10.1016/j.jclepro.2018.05.068
- [Background] Lange, F., & Dewitte, S. (2019). Measuring pro-environmental behavior: Review and recommendations. Journal of Environmental Psychology, 63, 92-100. https://doi.org/10.1016/j.jenvp.2019.04.009
- [Background] Loef M, Walach H. The combined effects of healthy lifestyle behaviors on all cause mortality: a systematic review and meta-analysis. Prev Med. 2012 Sep;55(3):163-70. doi: 10.1016/j.ypmed.2012.06.017. Epub 2012 Jun 24. PMID 22735042
- [Background] Mauch CE, Edney SM, Viana JNM, Gondalia S, Sellak H, Boud SJ, Nixon DD, Ryan JC. Precision health in behaviour change interventions: A scoping review. Prev Med. 2022 Oct;163:107192. doi: 10.1016/j.ypmed.2022.107192. Epub 2022 Aug 11. PMID 35963310
- [Background] Meader N, King K, Wright K, Graham HM, Petticrew M, Power C, White M, Sowden AJ. Multiple Risk Behavior Interventions: Meta-analyses of RCTs. Am J Prev Med. 2017 Jul;53(1):e19-e30. doi: 10.1016/j.amepre.2017.01.032. Epub 2017 Feb 28. PMID 28258777
- [Background] Moran, D., Wood, R., Hertwich, E., Mattson, K., Rodriguez, J. F. D., Schanes, K., & Barrett, J. (2020). Quantifying the potential for consumer-oriented policy to reduce European and foreign carbon emissions. Climate Policy, 20(sup1), S28-S38.
- [Background] Nisa CF, Belanger JJ, Schumpe BM, Faller DG. Meta-analysis of randomised controlled trials testing behavioural interventions to promote household action on climate change. Nat Commun. 2019 Oct 4;10(1):4545. doi: 10.1038/s41467-019-12457-2. PMID 31586060
- [Background] Nisbet, E. K. L., & Gick, M. L. (2008). Can health psychology help the planet? Applying theory and models of health behaviour to environmental actions. Canadian Psychology / Psychologie Canadienne, 49(4), 296-303.
- [Background] Osbaldiston, R., & Schott, J. P. (2012). Environmental Sustainability and Behavioral Science: Meta-Analysis of Proenvironmental Behavior Experiments. Environment and Behavior, 44(2), 257-299.
- [Background] Prochaska JJ, Spring B, Nigg CR. Multiple health behavior change research: an introduction and overview. Prev Med. 2008 Mar;46(3):181-8. doi: 10.1016/j.ypmed.2008.02.001. Epub 2008 Feb 6. PMID 18319098
- [Background] Riediger M, Freund AM. Interference and facilitation among personal goals: differential associations with subjective well-being and persistent goal pursuit. Pers Soc Psychol Bull. 2004 Dec;30(12):1511-23. doi: 10.1177/0146167204271184. PMID 15536236
- [Background] Santos, O., Virgolino, A., Vaz Carneiro, A., & De Matos, M. G. (2021). Health Behavior and Planetary Health: A Multi-Level Environmental Health Approach. European Psychologist, 26(3), 212-218.
- [Background] Steg, L., & Vlek, C. (2009). Encouraging pro-environmental behaviour: An integrative review and research agenda. Journal of Environmental Psychology, 29(3), 309-317.
- [Background] Truelove, H. B., Carrico, A. R., Weber, E. U., Raimi, K. T., & Vandenbergh, M. P. (2014). Positive and negative spillover of pro-environmental behavior: An integrative review and theoretical framework. Global Environmental Change, 29, 127-138.
- [Background] United Nations Development Programme. (2022). United Nations (UN).
- [Background] World Health Organization. COP26 special report on climate change and health: The health argument for climate action. Report No.: 9240036725. (2021). World Health Organization.
- [Background] Wu S, Zhu W, Thompson P, Hannun YA. Evaluating intrinsic and non-intrinsic cancer risk factors. Nat Commun. 2018 Aug 28;9(1):3490. doi: 10.1038/s41467-018-05467-z. PMID 30154431